CLINICAL TRIAL: NCT04267367
Title: Effectiveness of Dietitian-led Dietary Approach to Management of Diabetes (DIAM-D) in Tertiary Care Hospital of Nepal: a Randomized Control Trial
Brief Title: Effectiveness of Dietitian-led Dietary Approach to Management of Diabetes (DIAM-D)
Acronym: DIAM-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purbanchal University (Other)
Responsible Party: Principal Investigator, Devendra Raj Singh, Assistant Professor, Purbanchal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PurbanchalU
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Diabetes
Keywords: Dietitian; Dietary approach; Management; Diabetes; Nepal
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The source of the population of the study in both intervention and control group will be known cases of T2DM and newly diagnosed cases of T2DM patients who are within 20-64 years of age group attending the OPD of the hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will include a dietitian-led nutrition education, counseling session and individual basis diet plan emphasis on glycemic control diet targeted to T2DM patients attending during the OPD visits in hospital.
  Interventions: Behavioral: Dietitian-led dietary approach to management of diabetes
- Usual care (No Intervention): The usual care arm will be only provided general education.

INTERVENTIONS:
Behavioral: Dietitian-led dietary approach to management of diabetes — In the intervention phase, the educational and diet plan package will be developed. All the intervention packages will be approved by a multi-disciplinary expert team comprising an endocrinologist and dietitian prior to the intervention. Patients in the usual care arm will receive routine care as to how he/she is practicing in their daily life. Routine care includes general knowledge on diabetes disease process, blood glucose monitoring, a healthy lifestyle, preventing treating diabetes complications and developing personalized strategies for the decision-making process[27]. The intervention package will include mainly two-phase, nutritional counseling emphasis on lifestyle modification of diabetes patients and individual basis diet plan for each T2DM patients for intervention arm. The nutrition education and counseling and individual diet plan will be applied by trained dietitians.
  Arms: Intervention

SUMMARY:
Background: Diabetes mellitus is one of the major intractable public health problems in developing countries including Nepal. The dietary approach is of paramount significance in the management of type 2 diabetes. The nutrition education and counseling (NEC) may be good strategies for the management of diabetes provided by dietitians. There is still a lack of evidence on a dietitian-led dietary approach to the management of T2DM patients in the Nepalese context. The aims of this study is to examine the effectiveness of dietitian-led dietary approach to management of diabetes on reduction of HbA1c level, nutrition education score and macronutrient intake among T2DM patients in a tertiary care hospital in Kathmandu, Nepal.

Methods: The Dietary Approach to the Management of Diabetes (DIAM-D) trial is a hospital-based, open-label, two-armed, randomized control trial. A total of 156 participants with T2DM having HbA1c >6.5% will be enrolled in the study. Participants will be consecutively enrolled and assigned to receive nutrition education and counseling (NEC) and diet plan in the intervention group (n=78) and usual routine care in the control group (n=78) randomly. The NEC will be provided to participants on group session and the diet plan will be face-to-face individual basis at the time of enrollment and follow-ups will be done every month. Baseline data will be collected using a structured questionnaire for an interview and the biochemical tests will be measured. Baseline data will be collected at the time of enrollment, midline in three months and end-line data collection in 6 months. The primary outcome of the study will be a difference in mean change (from baseline, midline to 6 months) in the HbA1c level between the two study arms from baseline to end line. The secondary outcomes measure will be changed in biochemical and clinical parameters between the two arms at baseline midline to six months. Data will be entered using Epidata Software and transferred to the STATA/MP version 14.1 for further analysis. Data will be analyzed using an intention-to-treat basis. Independent sampele t-test and difference in the difference (DID) models will be used to estimates changes between the intervention and usual care arms.

DETAILED DESCRIPTION:
Background:

Diabetes mellitus (DM) refers to the metabolic syndrome characterized by high blood glucose levels considering major public health problems globally (Sun et al., 2018). The global prevalence of diabetes in adults has been increasing over the decades (Guariguata et al., 2014). According to the world health organization (WHO), diabetes is the sixth leading cause of death accounting for 1.59 million deaths in 2016 (World Health Organization (WHO)., 2018). According to the International Diabetes Federation (IDF) data, it was estimated that among 18-99 years, there are 451 million people with diabetes globally. The number projected to increase to 693 million by 2045 (Cho et al., 2018). The rapid change of diabetes prevalence in many countries specially developing countries have been influenced by rapid urbanization and drastically changes towards the sedentary lifestyle(Guariguata et al., 2014). Similarly, an increase in the prevalence of diabetes is characterized by various modifiable and non-modifiable risk factors, modifiable risk factors include changes in dietary habits and sedentary lifestyle which contributed to overweight/ obesity and non-modifiable risk factors including genetic cause and age (Hussain, Claussen, Ramachandran, & Williams, 2007).

The prevalence of diabetes mellitus in the south Asian region was a rapid increase over the last two decades (R.Jayawardena et al., 2012). According to the International Diabetes Federation (IDF) data for Nepal, the prevalence of T2DM in the 20-79 years age group was 4% in 2017 and the predicted number of undiagnosed cases was 532,100. IDF estimates the prevalence projected to increase by 6.1% and 1,264,200 undiagnosed cases in 2045 in Nepal(IDF Diabetes Atlas 9th edition 2019, n.d.). Evidence from systematic review and meta-analysis done by Gyawali et al, (2014) also reported that the prevalence of diabetes is a major public health problem with a prevalence rate of 8.4% (Gyawali et al., 2015). Dhimal et al. conducted a nationwide cross-sectional population-based study carried out from 2016-1018 found that the prevalence of diabetes was 8.5%(Dhimal et al., 2019). Diabetes is the third most common non-communicable disease in Nepal, which causes 12% of all hospitalizations(Bhandari, Angdembe, Dhimal, Neupane, & Bhusal, 2014).

Problem Statement:

The prevalence of type 2 diabetes mellitus (T2DM) has drastically increased in recent years in Nepal(Kafle, Poudel, & Shrestha, 2018). T2DM is accompanied by complications such as dyslipidemia, hypertension, and obesity. Several studies have shown that these complications can be prevented if lowering the HbA1c level and which has to be maintained within normal limits(Lim, Park, Choi, Huh, & Kim, 2009).

Dietary management is considered as the cornerstone of blood glucose level control in T2DM patients(Forouhi, Misra, Mohan, Taylor, & Yancy, 2018). Nowadays, nutrition education and counseling are the widely accepted strategies for the management of diabetes(Zheng, Liu, Liu, & Deng, 2019). Various studies have shown that T2DM patients are an association with nutrition education and improving dietary habits, nutritional knowledge and improving clinical outcomes such as lower blood glucose and HbA1c levels(Forouhi et al., 2018; Norris, Engelgau, & Narayan, 2001; Zheng et al., 2019). Once the diagnosis is confirmed to T2DM, patients are managed by mainly three approaches such as diet alone, diet and drugs or diet and insulin(Mbhenyanea, 2017). Indeed, dietary factors are crucial for the management and prevention of T2DM (Forouhi et al., 2018). Furthermore, individualized nutrition education and counseling are effective strategies in adherence to diet recommendations and in improving glycemic control(Lim et al., 2009). Dietitian-led nutrition education and lifestyle intervention are effective in reducing body weight and glucose-related outcomes(Sun et al., 2018). However, limited studies have been carried out to examine the effectiveness of a dietary approach to the management of diabetes consulted by a dietitian in developing countries (Huang, Hsu, Wang, & Shin, 2010; Trento et al., 2008). Therefore, there is still a lack of evidence on effective guidelines and protocols for a dietitian-led dietary approach to the prevention and management of T2DM patients.

Literature Review and Research Gaps:

Diabetes is one of the major public health problems globally with projected to increase the estimated prevalence is 425 million people in 2017 to 629 million by 2045(Forouhi et al., 2018). Most of the developing countries including Nepal are experienced and increasing the burden of non-communicable diseases such as diabetes mellitus(Gyawali et al., 2015). A recently published study showed 8.5% of peoples have diabetes in the context of Nepal with 5.5% living in rural areas and higher peoples 11.3% are living in urban areas(Nepal Health Research Council, 2019).

In the context of Nepal, most of the peoples are tend to consume a diet rich in simple sugar-containing foods rather than complex carbohydrate and dietary fiber and sedentary lifestyle resulting greatly increased the levels of lifestyle-related disease such as diabetes(Hills et al., 2018). Thus, changing dietary habits can shift a society's disease pattern from infectious, communicable diseases' dominance towards a status of double-burden disease with an increasing prevalence of obesity and non-communicable diseases (NCDs) such as diabetes mellitus(Bishwajit, 2015). Evidence from high-income countries (HICs) shows that healthy eating habits and dietary guidelines area good strategies for the management of diabetes(Forouhi et al., 2018). Therefore, the government of Nepal now prioritizes health promotion for NCDs(Ministry of Health and Population., 2015).

Dietitians can play an important role in the management of non-communicable diseases such as diabetes through nutritional counseling and dietary modification. Nowadays, the provision of nutritional counseling and individualized diet plan concept consulted by dietitians has been practicing in most of the hospital in Nepal. However, there is still lacking the evidence-based dietary guidelines in the Nepalese context. To our knowledge, the effectiveness of the management of diabetes consulted by dietitians has not been explored yet in Nepal. The investigators intended to examine the effectiveness of a dietitian-led dietary approach to management for diabetes mellitus among T2DM patients in tertiary care hospitals. The investigators also tried to examine the future direction for effective dietary and nutritional management approaches to manage T2DM and their implementation in the Nepalese context. Eventually, these outcomes of the study will bridge the evidence gap regarding the scope and provision of dietitians in every government and non-government hospital to the prevention and management of non-communicable diseases such as T2DM.

Research hypothesis:

Dietitian-led dietary approach to the management of diabetes will improve on HbA1c level, nutrition knowledge score and macronutrient intake level compared to usual care among type 2 diabetes mellitus patients in tertiary care hospital in Nepal.

General objectives :

The main objective of this study is to evaluate the effectiveness of the dietitian-led dietary approach to the management of diabetes on the reduction of HbA1c level, nutrition education score and macronutrient intake among T2DM patients in a tertiary care hospital in Kathmandu, Nepal.

Specific objectives :

To measure the change in HbA1c level among T2DM patients between the intervention and control/usual care arm.

To evaluate the change in macronutrient intake level among T2DM patients in the intervention and usual care arm.

To assess dietitian-led nutrition education and counseling on nutritional knowledge of diabetes among T2DM patients.

To evaluate the change in biochemical parameters among T2DM patients in the intervention and usual care arm.

To assess the nutritional status such as BMI and WHR among T2DM patients

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of type 2 diabetes with (as defined by an HbA1c>48 mmol/mol (6.5%) at time of diagnosis)
* Male or female aged ≥20 years and visited in OPD of target hospital
* Those who give consent to participate in our intervention study

Exclusion Criteria:

* Those who are pregnant women, lactating women or planning to become pregnant during the course of study.
* Those who are severely ill or more than two comorbidities
* Those who have any plan to migrate from the study area for at least 1 year
* HbA1c ≥93mmol/mol (10.5%)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level | six months
  The primary outcome of this study will be the change in mean HbA1c between the intervention and control/usual care groups from baseline to end line.

CONTACTS AND LOCATIONS:
Overall Officials: Devendra Raj Singh, MScHPPH, Principal Investigator — Asian College for Advance Studies, Purbanchal University
Locations (1):
- Asian College for Advance Studies, Purbanchal University, Lalitpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forouhi NG, Misra A, Mohan V, Taylor R, Yancy W. Dietary and nutritional approaches for prevention and management of type 2 diabetes. BMJ. 2018 Jun 13;361:k2234. doi: 10.1136/bmj.k2234. PMID 29898883
- [Result] Sun Y, You W, Almeida F, Estabrooks P, Davy B. The Effectiveness and Cost of Lifestyle Interventions Including Nutrition Education for Diabetes Prevention: A Systematic Review and Meta-Analysis. J Acad Nutr Diet. 2017 Mar;117(3):404-421.e36. doi: 10.1016/j.jand.2016.11.016. PMID 28236962
- [Result] Guariguata L, Whiting DR, Hambleton I, Beagley J, Linnenkamp U, Shaw JE. Global estimates of diabetes prevalence for 2013 and projections for 2035. Diabetes Res Clin Pract. 2014 Feb;103(2):137-49. doi: 10.1016/j.diabres.2013.11.002. Epub 2013 Dec 1. PMID 24630390
- [Result] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Result] Jayawardena R, Ranasinghe P, Byrne NM, Soares MJ, Katulanda P, Hills AP. Prevalence and trends of the diabetes epidemic in South Asia: a systematic review and meta-analysis. BMC Public Health. 2012 May 25;12:380. doi: 10.1186/1471-2458-12-380. PMID 22630043
- [Result] Gyawali B, Sharma R, Neupane D, Mishra SR, van Teijlingen E, Kallestrup P. Prevalence of type 2 diabetes in Nepal: a systematic review and meta-analysis from 2000 to 2014. Glob Health Action. 2015 Nov 26;8:29088. doi: 10.3402/gha.v8.29088. eCollection 2015. PMID 26613684
- [Result] Lim HM, Park JE, Choi YJ, Huh KB, Kim WY. Individualized diabetes nutrition education improves compliance with diet prescription. Nutr Res Pract. 2009 Winter;3(4):315-22. doi: 10.4162/nrp.2009.3.4.315. Epub 2009 Dec 31. PMID 20098585
- [Result] Bhandari GP, Angdembe MR, Dhimal M, Neupane S, Bhusal C. State of non-communicable diseases in Nepal. BMC Public Health. 2014 Jan 10;14:23. doi: 10.1186/1471-2458-14-23. PMID 24405646
- [Result] Zheng F, Liu S, Liu Y, Deng L. Effects of an Outpatient Diabetes Self-Management Education on Patients with Type 2 Diabetes in China: A Randomized Controlled Trial. J Diabetes Res. 2019 Jan 17;2019:1073131. doi: 10.1155/2019/1073131. eCollection 2019. PMID 30800684
- [Result] Bishwajit G. Nutrition transition in South Asia: the emergence of non-communicable chronic diseases. F1000Res. 2015 Jan 12;4:8. doi: 10.12688/f1000research.5732.2. eCollection 2015. PMID 26834976
- [Result] Dhimal M, Karki KB, Sharma SK, Aryal KK, Shrestha N, Poudyal A, Mahato NK, Karakheti A, Sijapati MJ, Khanal PR, Mehata S, Vaidya A, Yadav BK, Adhikary KP, Jha AK. Prevalence of Selected Chronic Non-Communicable Diseases in Nepal. J Nepal Health Res Counc. 2019 Nov 14;17(3):394-401. doi: 10.33314/jnhrc.v17i3.2327. PMID 31735938
- [Derived] Sunuwar DR, Nayaju S, Dhungana RR, Karki K, Singh Pradhan PM, Poudel P, Nepal C, Thapa M, Shakya NS, Sayami M, Shrestha PK, Yadav R, Singh DR. Effectiveness of a dietician-led intervention in reducing glycated haemoglobin among people with type 2 diabetes in Nepal: a single centre, open-label, randomised controlled trial. Lancet Reg Health Southeast Asia. 2023 Sep 25;18:100285. doi: 10.1016/j.lansea.2023.100285. eCollection 2023 Nov. PMID 38028163
- See also: World Health Organization (WHO). The top 10 causes of death. 2018. — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death
- See also: Kafle N, Poudel R, Shrestha S. Noncompliance to Diet and Medication among Patients with Type 2 Diabetes Mellitus in Selected Hospitals of Kathmandu, Nepal. J Soc Heal Diabetes. — http://www.thieme-connect.com/products/ejournals/pdf/10.1055/s-0038-1675687.pdf
- See also: Nepal Health Research Council. Population Based Prevalence of Selected Non-Communicable Disease in Nepal. 2019. — http://www.ghbook.ir/index.php?namecom_
- See also: Ministry of Health and Population. Nepal Health Sector Strategy 2015-2020, Kathmandu. 2015. — https://www.healthynewbornnetwork.org/hnn-content/uploads/NHSS_English_Book.pdf